CLINICAL TRIAL: NCT06525116
Title: Measurable Residual Disease Detection by Next-generation Sequencing of T Cell Receptor Gene Rearrangements in Pediatric T-cell Acute Lymphocytic Leukemia
Brief Title: MRD Detection by NGS in Pediatric T-ALL
Status: Completed | Type: Observational
Sponsor: The Children's Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Principal Investigator, Xiaojun Xu, Principal investigator, The Children's Hospital of Zhejiang University School of Medicine
Other Study IDs: 2024-IRB-0210-P-01
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Acute Lymphoblastic Leukemia, Pediatric
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MRD — Calculate the 3-year EFS based on the MRD status (MRD positive and negative groups)

SUMMARY:
This retrospective analysis aims to investigate pediatric patients with T cell acute lymphoblastic leukemia who were detected for minimal residual disease (MRD) using next-generation sequencing (NGS). The study will utilize second-generation sequencing technology to analyze the rearrangement of the T cell receptor (TCR) genes in these patients. Patients will be stratified based on NGS-MRD levels, and the relationship between NGS MRD and Event-Free Survival (EFS) will be evaluated.

DETAILED DESCRIPTION:
This was a prospective, single-center, observational study conducted in children with ALL between February 2018 and December 2022. Children with newly diagnosed T-ALL who undergone NGS of T-cell receptors at Children's Hospital，Zhejiang University School of Medicine were included in this study. The European Group for the Immunological Characterization of Leukemias (EGIL) criteria were applied to diagnose and classify ALL in this study. All enrolled patients were treated according to the ZJCH-ALL-2019 protocol detailed in the supplementary file. This protocol was implemented in our center in September 2018 and subsequently extended to all of Zhejiang Province in 2019. In this protocol, NGS-MRD was not used for patient risk stratification or treatment allocation. For the detection of MRD, bone marrow (BM) aspiration for NGS was collected at diagnosis. Multiple consecutive MRD test evaluation points (TP) were set up, including but not limited to at least day 15 of induction remission, the end of induction remission (EOI), the end of consolidation therapy (EOC), 6 months after diagnosis (6-month). NGS-MRD was sequentially monitored every 3 to 6 months after EOC until it was undetectable. In this study, NGS-MRD refers to the quantitative value of MRD detected through NGS testing which was the sum of TRB/TRG levels. The patients were followed up until June 30, 2024. Statistical Analysis The association between categorical variables was tested using χ2 test, the correlation between quantitative variables was measured using Pearson correlation and tested using Student's t distribution, and ANOVA was used to compare quantitative variables. Event-free survival (EFS) and overall survival (OS) curves were estimated using the Kaplan-Meier method and compared according to the log rank test. Death during induction, abandonment before complete remission, death in continuous complete remission, relapse, and secondary malignancies were considered as events in the calculation of EFS probability. The EFS time was calculated from the date of diagnosis to the last date of follow-up or the first event. The OS was calculated from the date of diagnosis to death from any causes with censoring the patients alive at the time of data analysis. Data visualization was performed using R package ggplot2 (Version 4.0.3) and GraphPad Prism 8.0.0. Statistical analysis was performed on R (Version 4.0.3). A P value <0.05 (two tailed) was considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Children with newly diagnosed T-ALL who undergone NGS of T-cell receptors

Exclusion Criteria:

* T-ALL patients who have not undergone high-throughput sequencing.
* T-ALL Patients without traceable significant clones.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children under the age of 18 years diagnosed with acute T-cell lymphoblastic leukemia between 2018 and 2022
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
event-free survival | Between February 2018 and December 2022
  The EFS time was calculated from the date of diagnosis to the last date of follow-up or the first event.

CONTACTS AND LOCATIONS:
Locations (1):
- The Children's Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China